CLINICAL TRIAL: NCT00522054
Title: Tai Chi for Patients With Rheumatoid Arthritis: A Quantitative and Qualitative Study
Brief Title: Tai Chi for Patients With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 587-03244
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2007-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Exercise; Physical function; Rheumatoid arthritis; Tai Chi
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): Single group study
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — Tai Chi exercise, twice a week during 12 weeks

SUMMARY:
The purpose of this study was to study the impact of Tai Chi group exercise on physical function, health and disease activity of patients with RA, and to examine the patients' experience and perception of Tai Chi.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic, inflammatory and systemic disease that mainly affects the musculoskeletal system. The disease is often progressive and may result in reduced physical function, pain, fatigue, and joint destruction. Exercise programs are reported to improve physical functioning in patients with RA.

Tai Chi is a traditional Chinese martial art that was developed in the 13th century, and combines slow and gentle movements with mental focus.

The aim of this study was to examine the impact of a 12 weeks standardized Tai Chi group exercise program on disease activity, physical function and health status in patients with RA attending. Further, the patients experiences of possible effects of Tai Chi were to be obtained in a focus group interview.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA according to the American College of Rheumatology (ACR) 1987
* Stable medical treatment
* No earlier experience with Tai Chi

Exclusion Criteria:

* Lack of ability to bear weight on the lower extremities
* Recent or ongoing disease flare
* Unstable heart condition
* Participation in other physical exercise interventions more than twice a week included in other intervention studies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-09; Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Balance was measured with Walking in a Figure of Eight. Strength and endurance were measured by Timed-Stands test. Shoulder function was measured with Assessments of Shoulder Movement Impairment Scale. | 15 min

SECONDARY OUTCOMES:
Blood samples were collected for determination of sedimentation rate (ESR) and C-reactive protein (CRP). A rheumatologist examined the patients with the number of 28 swollen and tender joints. | 15 min
Self-reported health status included Health Assessment Questionnaire, visual analogue scale for fatigue, muscle pain, and fear of falling, Short Form Health Survey and Arthritis Self-Efficacy Scale | 15 min
Focus group interview in order to capture the participants' experiences and perceptions with Tai Chi. | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Fongen, MSc, Study Chair — National Resource Center for Rehabilitation in Rheumatology
Locations (1):
- National resource center for rehabilitation in rheumatology. Diakonhjemmet Hospital, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Uhlig T, Fongen C, Steen E, Christie A, Odegard S. Exploring Tai Chi in rheumatoid arthritis: a quantitative and qualitative study. BMC Musculoskelet Disord. 2010 Mar 5;11:43. doi: 10.1186/1471-2474-11-43. PMID 20205741